CLINICAL TRIAL: NCT01345305
Title: Establishing Reliability for Quantitative EEG, Transcranial Doppler, Behavioral Outcomes and Optical Coherence Tomography in SWS: The Next Step Toward Biomarker Development
Brief Title: Biomarker Development in Sturge-Weber Syndrome
Acronym: Pilot
Status: Completed | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of California, San Francisco (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Anne Comi, MD, Associate Professor, Neurology and Developmental Medicine, Kennedy Krieger Institute, Johns Hopkins University, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Other Study IDs: NA_00043846; BVMC6204 (Other: Rare Diseases Clinical Research Network); U54NS065705-02 (NIH)
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Sturge-Weber Syndrome
Keywords: Sturge-Weber Syndrome; Biomarkers; Quantitative EEG; Transcranial Doppler Ultrasound; Medical Rehabilitation Scales; Optical Coherence Tomography
MeSH Terms: conditions — Sturge-Weber Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study of 40 individuals with Sturge-Weber Syndrome (SWS) brain and/or eye involvement. It will examine the test-retest reliability of the following clinical tests:

1. Quantitative EEG
2. Transcranial Doppler
3. Medical Rehabilitation Scales
4. Optical Coherence Tomography

DETAILED DESCRIPTION:
Sturge-Weber Syndrome (SWS) is a rare disorder presenting at birth with a facial port-wine birthmark and later in infancy with seizures and strokes that result in weakness on one side of the body, cognitive disabilities, glaucoma, and visual field deficits. Approximately 10-50% of infants born with a facial port-wine birthmark on the upper part of the face will also have SWS brain and/or eye involvement. Early detection and treatment of the disease is necessary to improve an SWS patient's outcome, and early biological indicators need to be discovered to make this possible. We believe the following tests can serve as non-invasive biomarkers to improve early diagnosis, monitor response to treatment, and to predict outcome:

1. Quantitative EEG
2. Transcranial Doppler
3. Medical Rehabilitation Scales
4. Optical Coherence Tomography The first step of this process is to determine how much the results of these tests vary between individual tests.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with SWS and brain involvement (Aims 1-3): for the purposes of this study SWS brain involvement is defined as having shown on MRI imaging evidence of the typical vascular malformation which includes the following: leptomeningeal angioma, choroid plexus glomus, and associated venous angioma/malformation.
2. Individuals with SWS and eye involvement (Aim 4): for the purposes of this study SWS eye involvement is defined as individuals with a port-wine birthmark in the V1 dermatomal distribution
3. Able (or parents able) to provide informed consent
4. Able to cooperate with tests
5. Age 6 months to 21 years (Aims 1-3 only)

Exclusion Criteria:

* Subjects unable to cooperate with the studies will be excluded.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Individuals with SWS and brain involvement (Aims 1-3): for the purposes of this study SWS brain involvement is defined as having shown on MRI imaging evidence of the typical vascular malformation which includes the following: leptomeningeal angioma, choroid plexus glomus, and associated venous angioma/malformation.
  2. Individuals with SWS and eye involvement (Aim 4): for the purposes of this study SWS eye involvement is defined as individuals with a portwine birthmark in the V1 dermatomal distribution
  3. Able (or parents able) to provide informed consent
  4. Able to cooperate with tests
  5. Age 6 months to 21 years (Aims 1-3 only)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 2 years
  Our primary aim is to demonstrate correlation between progression of clinical symptoms and evolution of the vascular malformation involving the brain, skin, and the eye.

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Comi, M.D., Principal Investigator — Hunter Nelson Sturge-Weber Center
Locations (1):
- Hunter Nelson Sturge-Weber Center at Kennedy Krieger Institute, Baltimore, Maryland, United States